CLINICAL TRIAL: NCT02024490
Title: The Effect of Maternal and Neonatal Vitamin D Levels on Respiratory Distress Syndrome in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merih Cetinkaya, Associate Professor, MD, PhD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: MC10001
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D, prematurity, RDS, BPD, maternal, neonatal
MeSH Terms: conditions — Vitamin D Deficiency; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RDS group, non-RDS group: RDS group; infants with clinical, radiological and laboratory findings of RDS non-RDS group; infants without clinical, radiological and laboratory findings of RDS

SUMMARY:
Respiratory distress syndrome (RDS) of the newborn, also called as hyaline membrane disease, is the most common cause of respiratory distress in premature infants, correlating with structural and functional lung immaturity. The pathophysiology of RDS is complex. Immature type II alveolar cells produce less surfactant that causes an increase in alveolar surface tension and a decrease in compliance. This resultant atelectasis lead to pulmonary vascular constriction, hypoperfusion, and lung tissue ischemia. RDS and prolonged ventilation and associated systemic/lung injury may also contribute to long term oxygen dependency and may result in bronchopulmonary dysplasia (BPD). Vitamin D is a fat-soluble steroid hormone that primarily contributes to the maintenance of normal calcium homeostasis and skeletal mineralization. In addition to its classical role in bone metabolism, vitamin D deficiency has been associated with impaired pulmonary function, increased incidence of viral and bacterial infections and inflammatory lung diseases. Although exact mechanisms are not fully understood, vitamin D appears to impact on a variety of inflammatory and structural cells within the lung including macrophages, lymphocytes and epithelial cells. To our best of knowledge, no study has evaluated the effect of vitamin D levels on the severity and presence of RDS in preterm infants. Therefore, the aim of this study is to evaluate the possible role of maternal/neonatal vitamin D levels on RDS development in preterm infants. We also aim to determine the possible association between maternal/neonatal vitamin D levels and the incidence of BPD and other neonatal morbidities.

DETAILED DESCRIPTION:
Preterm infants with respiratory distress who are <37 weeks of gestational age and will be admitted to Neonatal Intensive Care Unit of Kanuni Sultan Suleyman Training and Research Hospital will be included in this prospective study. Blood for neonatal and maternal vitamin D levels will be obtained from all infants and their mothers at the time of hospital admission. The infants will be evaluated for RDS and surfactant requirement. If they have RDS and need of mechanical ventilation, they will be intubated and given surfactant, if necessary. The maternal and neonatal demographics of infants will be recorded. Infants will also be followed up in terms of other morbidities including patent ductus arteriosus, necrotizing enterocolitis, retinopathy of prematurity, and especially BPD. Then infants will be divided into three groups according to maternal/neonatal vitamin D levels (mild, moderate and severe vitamin D deficiency) and group comparisons will be performed Plasmas after separated and stored at -80 C. Levels of 25-OHD will be determined using Shimadzu LC-20AT model High Performance Liquid Chromatography (HPLC) system. Data will be analyzed using SPSS software and appropriate statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <37 weeks of gestational age and are admitted to Neonatal Intensive Care Unit of Kanuni Sultan Suleyman Training and Research Hospital
* Preterm infants with clinical and laboratory findings of RDS

Exclusion Criteria:

* presence of maternal clinical and/or histological chorioamnionitis,
* presence of premature rupture of membranes (PROM),
* refusal of parental consent,
* lack of laboratory data,
* major congenital abnormalities

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants admitted to neonatal intesive care unit with the diagnosis of respiratory distress syndrome (RDS) will constitute the RDS group, whereas preterm infants without RDS will constitute the non-RDS group
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
development of respiratory distress in infants according to vitamin D levels | 1 year
  A total of 100 preterm infants will be included and vitamin D levels will be compared between those with and without respiratory distress syndrome

SECONDARY OUTCOMES:
presence of vitamin D deficiency and bronchopulmonary dysplasia | 1 year

OTHER OUTCOMES:
development of prematurity morbidities | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Merih Cetinkaya, MD, PhD, Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Stanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Parekh D, Thickett DR, Turner AM. Vitamin D deficiency and acute lung injury. Inflamm Allergy Drug Targets. 2013 Aug;12(4):253-61. doi: 10.2174/18715281113129990049. PMID 23782208
- [Background] Gupta A, Bush A, Hawrylowicz C, Saglani S. Vitamin D and asthma in children. Paediatr Respir Rev. 2012 Dec;13(4):236-43; quiz 243. doi: 10.1016/j.prrv.2011.07.003. Epub 2011 Sep 1. PMID 23069123
- [Background] Bener A, Ehlayel MS, Tulic MK, Hamid Q. Vitamin D deficiency as a strong predictor of asthma in children. Int Arch Allergy Immunol. 2012;157(2):168-75. doi: 10.1159/000323941. Epub 2011 Oct 6. PMID 21986034